CLINICAL TRIAL: NCT05608486
Title: Continuation Protocol for Study Using Negative Pressure to Reduce Apnea Trial (CO-STAR)
Brief Title: Continuation Protocol for Study Using Negative Pressure to Reduce Apnea Trial
Acronym: CO-STAR
Status: Available | Type: Expanded Access
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SOM-030
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

INTERVENTIONS:
Device: aerSleep II — The aerSleep® II System includes a soft silicone collar, which is placed on the anterior neck. Integrated with the collar is a vacuum pump module (VPM), which cordlessly powers the generation of negative pressure within the collar's cavity. This negative pressure pulls the underlying tissues forward, maintaining airway patency.
  Other Names: Continuous Negative External Pressure (cNEP)

SUMMARY:
The goal of this study is to allow continued access to the aerSleep II System for subjects that have completed the SOM-029 study until the device is commercially available.

DETAILED DESCRIPTION:
This is a multi-center uncontrolled continuation study designed to mimic real-world use of the aerSleep II System for subjects that have completed the SOM-029 protocol.

Subjects will use the aerSleep II nightly at a fixed pressure of -30 cmH2O. Internal electronics will record various measures of how the device is being used and how it performs.

Subjects will have a video visit with the study site approximately every 30 days, and, if the Investigator feels it is warranted or at the subject's discretion, an in-person visit at the study site will occur approximately every 90 days. During these visits, subjects will be queried for adverse events and asked to complete simple subjective evaluations of their experiences. The Investigator will complete a scale rating how well the device is managing the subject's obstructive sleep apnea (OSA).

Data collected from the device will be retrieved approximately every 90 days to monitor vacuum delivery and subject compliance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject completed study SOM-029 (SUPRA).
2. The Investigator feels that the subject experienced sufficient benefit from aerSleep II to justify its further use.
3. In the Investigator's judgement, the subject will be able to understand and comply with all study procedures.

Exclusion Criteria:

1. The Investigator feels that, for any reason, the subject's participation may not be in his or her best interest.
2. Any condition or circumstance that in the opinion of the Investigator is likely to prevent accurate data collection or bias the results.
3. The subject is pregnant or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kingman P. Strohl, M.D., Principal Investigator — Case Western Reserve University School of Medicine